CLINICAL TRIAL: NCT04077580
Title: The Effect of Methenamine Hippurate to Reduce Antibiotic Prescribing Due to New Episodes of Urinary Tract Infections (UTI) in Elderly Women With Recurrent UTI - a Triple- Blinded, Randomized Placebo-controlled Phase IV Study
Brief Title: The Effect of Methenamine Hippurate to Reduce Antibiotic Prescribing in Elderly Women With Recurrent UTI
Acronym: ImpresUWP3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); UMC Utrecht (Other); Göteborg University (Other); Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Morten Lindbaek, professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eudract 2018-002235-15
Record Dates: First submitted 2019-08-12; First posted 2019-09-04 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: blinded randomized trial; frail elderly women; prevention
MeSH Terms: conditions — Urinary Tract Infections | interventions — methenamine hippurate

STUDY DESIGN:
Intervention Model Description: We will perform a randomised trial in the targeted population, women >70 years in general practice in the 4 countries. Nursing home patients may be included, all shall give informed consent. Approximately 100 patients in each country.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomisation list will be generated by computer with individual randomisation. Kragerø Tablettproduksjon AS will pack and label IMP with active substance and placebo according to the randomisation list. Participants will be dispensed Investigational Medical Product (IMP) in consecutive order at each study site, through a designated pharmacy, one site in each country. Kragerø Tablettproduksjon AS will have the list available at all times with the possibility to break the code. In addition there will be one envelope for each medication identification (ID) available in each country, at the coordinating centres, containing information of active substance or placebo regarding IMP delivered to that specific country. These envelopes will be stored together with the IMP in a locker. In acute situations, the PI in each country will be able to break the code and disrupt the unblinding process without the consent of the sponsor in order not to hamper necessary medical treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methenamine hippurate (Experimental): Tablets containing 1 g methenamine hippurate, dosage 1 tablet morning and evening.
  Interventions: Drug: Methenamine Hippurate 1000 MG
- Placebo (Placebo Comparator): Placebo tablets containing 1 g of lactose, with identical size, shape and stamps
  Interventions: Drug: Methenamine Hippurate 1000 MG

INTERVENTIONS:
Drug: Methenamine Hippurate 1000 MG — Methenamine and placebo is taken 1 tablet morning and evening for 180 days
  Other Names: Placebo tablets with identical size, shape and stamps

SUMMARY:
Recurrent urinary tract infection (UTI) in elderly women is a major driver of antibiotic prescription. Hence, the question of feasible and appropriate preventive measures are important issues in this field. Methenamine hippurate is frequently prescribed in Norway and Sweden as prophylaxis for recurrent UTI. Methenamine hippurate acts via the production of formaldehyde from hexamine, which in turn acts as a bacteriostatic agent, therefore methenamine hippurate is not defined as an antibiotic. According to a Cochrane review 2012 the rates of adverse events for preventing UTI was low. Although this review showed methenamine hippurate might be effective in preventing UTI in the short term, there is a need for large well-conducted randomised controlled trial (RCT) to clarify both the safety and effectivity of preventive methenamine hippurate for longer term use. This is particularly important for longer term use for people without neuropathic bladder disorders. A Norwegian longitudinal observational study including women aged 50-80 years with recurrent UTI indicated a significant and large reduction of more than 50% in antibiotic prescriptions for UTI after start of prophylactic methenamine hippurate. This further strengthens the need for an RCT of methenamine hippurate as prophylaxis for recurrent UTI.

DETAILED DESCRIPTION:
Rationale for conducting this study:

Existing knowledge suggests that methenamine hippurate is a safe drug with few and mild side effects and with the potential to significantly reduce antibiotic usage for women with recurrent UTIs. Methenamine hippurate has been on the market for a long time but has never been tested to prevent recurrent UTIs in larger RCTs with long time follow-up. Hence, this must be proven in a large randomised trial before recommending large scale use of this drug.

The primary objective of this study is to investigate if taking methenamine hippurate reduce the need for antibiotic usage due to recurrent UTI (measured as number of antibiotic courses). Pyelonephritis, hospitalization and death will be registered as safety endpoints in the study.

Study design: Triple- blinded randomised controlled phase IV trial where patients are randomised to active intervention (methenamine hippurate) or controls (placebo). We will include women aged ≥ 70 years with recurrent UTIs, defined as ≥ 3 episodes of antibiotic treated acute cystitis (acute symptoms specific/related to the urinary tract) during the last twelve months or ≥ 2 episodes during the last six months.

Setting and study population:

Women aged ≥ 70 years with recurrent UTIs in primary care. A total of 400 patients will be randomized in this trial, with approximately 100 patients in each of the participating countries; Norway, Sweden, Poland and the Netherlands. The patients will be treated for 6 months.

Patients will be enrolled August-December 2019, including screening for eligibility and getting informed consent.

Start of study with drugs is from October 1st 2019.

Primary outcome: Number of UTI antibiotic treatments during the six months of treatment. If the participant receives >1 antibiotic courses for UTI without symptom relief it is regarded as one episode and counted as one antibiotic treatment. If there has been an asymptomatic period of at least 14 days in-between two UTI antibiotic courses, this is regarded as a new antibiotic treatment. Outcomes will be assessed after 6 and 12 months

In the analysis standard linear regression will be used where number of UTI antibiotic treatments will be the dependent variable. Group allocation together with the confounding variables above will be independent variables. The dependent variable will be transformed using a rank transformation in case it is not normally distributed. A p-value will be delivered but no useful effect size if a rank transformation is used.

ELIGIBILITY:
Inclusion Criteria:

* woman
* age ≥ 70 years
* recurrent UTIs defined as ≥ 3 episodes of antibiotic treated acute cystitis (acute symptoms specific/related to the urinary tract) during the last twelve months or ≥ 2 episodes during the last 6 months
* able and willing to comply with all trial requirements
* able and willing to give informed consent

Exclusion Criteria:

* the patient has taken methenamine hippurate within the last 12 months
* the patient is allergic to methenamine hippurate
* the patient is having current antibiotic prophylaxis for UTI
* the patient has a urinary catheter (chronic indwelling catheters as well as intermittent urinary catheterisation)
* the patient has known severe chronic renal failure or estimated creatinine glomerular filtration rate ≤ 30 ml/min (known = registered in general practice clinical records)
* the patient has a known condition or treatment associated with significant impaired immunity (e.g. long-term oral steroids, chemotherapy, or immune disorder) (known = registered in general practice (GP) clinical records)
* the patient has a known severe hepatic impairment (known = registered in GP clinical records)
* the patient is suffering from severe dehydration
* the patient has shown signs of gout
* the patient has a need for long term use of antacids such as magnesium hydroxide, magnesium carbonate, aluminium hydroxide
* the patient has a life expectancy estimated by a clinician to be less than six months
* the patient has been involved in, including completion of, follow-up procedures, in another clinical trial of an investigational medicinal product in the last 90 days
* the patient suffers from incontinence too severe to be able to provide a voided urine specimen
* the patient is participating in ImpresU Work Package 2
* the patient is suffering from significant known abnormal renal tract anatomy/physiology or neuropathic bladder disorders.
* The patient has intolerance versus lactose

Ages: 70 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 289 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate if taking methenamine hippurate reduces the need for antibiotic usage due to recurrent UTI (measured as number of antibiotic courses). | 6 months
  Number of UTI antibiotic treatments during the six months of treatment. If the participant receives >1 antibiotic courses for UTI without symptom relief it is regarded as one episode and counted as one antibiotic treatment. If there has been an asymptomatic period of at least 14 days in-between two UTI antibiotic courses, this is regarded as a new antibiotic treatment.

SECONDARY OUTCOMES:
Use of methenamine will give prolonged effect on antibiotic usage . | 6 months after stop of trial treatment
  Number of UTI antibiotic treatments during the six months following completion of treatment.
Use of methenamine will reduced incidence of UTI. | 6 months
  Number of UTIs (acute symptoms specific/related to the urinary tract) during the six months of treatment.
Use of methenamine reduce severity of UTI symptoms. | 6 months
  Registration of symptom severity when initiating treatment for UTI
Use of methenamine hippurate reduce duration of UTI episodes. | 6 months
  Registration of number of days of symptoms during UTI episodes.
Use of methenamine will reduce complications such as pyelonephritis and hospital admission for UTI | 6 months
  register complications such as pyelonephritis and hospital admission for UTI

CONTACTS AND LOCATIONS:
Overall Officials: Cees Hertogh, prof.MD, Principal Investigator — Amsterdam UMC, location VUmc; Theo Verheij, prof. MD, Principal Investigator — UMC Utrecht; Maciek Godycki.Cwirko, prof MD, Principal Investigator — Medical University of Lodz; Per-Daniel Sundvall, MD PhD, Principal Investigator — Vastra Gotaland Region
Locations (4):
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- University of Oslo, Oslo, Norway
- Medical University of Lodz,, Lodz, Poland
- Research and Development Primary Health Care, Region Västra Götaland,, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee BS, Bhuta T, Simpson JM, Craig JC. Methenamine hippurate for preventing urinary tract infections. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD003265. doi: 10.1002/14651858.CD003265.pub3. PMID 23076896
- [Result] Davis C, Rantell A. Lower urinary tract infections in women. Br J Nurs. 2017 May 11;26(9):S12-S19. doi: 10.12968/bjon.2017.26.9.S12. PMID 28493770
- [Result] Barclay J, Veeratterapillay R, Harding C. Non-antibiotic options for recurrent urinary tract infections in women. BMJ. 2017 Nov 23;359:j5193. doi: 10.1136/bmj.j5193. No abstract available. PMID 29170359
- [Result] Aydin A, Ahmed K, Zaman I, Khan MS, Dasgupta P. Recurrent urinary tract infections in women. Int Urogynecol J. 2015 Jun;26(6):795-804. doi: 10.1007/s00192-014-2569-5. Epub 2014 Nov 20. PMID 25410372
- [Result] van Buul LW, van der Steen JT, Veenhuizen RB, Achterberg WP, Schellevis FG, Essink RT, van Benthem BH, Natsch S, Hertogh CM. Antibiotic use and resistance in long term care facilities. J Am Med Dir Assoc. 2012 Jul;13(6):568.e1-13. doi: 10.1016/j.jamda.2012.04.004. Epub 2012 May 9. PMID 22575772
- [Result] Sundvall PD, Stuart B, Davis M, Roderick P, Moore M. Antibiotic use in the care home setting: a retrospective cohort study analysing routine data. BMC Geriatr. 2015 Jun 25;15:71. doi: 10.1186/s12877-015-0073-5. PMID 26108340
- [Result] Cronberg S, Welin CO, Henriksson L, Hellsten S, Persson KM, Stenberg P. Prevention of recurrent acute cystitis by methenamine hippurate: double blind controlled crossover long term study. Br Med J (Clin Res Ed). 1987 Jun 13;294(6586):1507-8. doi: 10.1136/bmj.294.6586.1507. PMID 3111615
- [Result] Brumfitt W, Hamilton-Miller JM, Gargan RA, Cooper J, Smith GW. Long-term prophylaxis of urinary infections in women: comparative trial of trimethoprim, methenamine hippurate and topical povidone-iodine. J Urol. 1983 Dec;130(6):1110-4. doi: 10.1016/s0022-5347(17)51709-7. PMID 6227756
- [Result] Alberg T, Holen O, Blix HS, Lindbaek M, Bentele H, Eriksen HM. Antibiotic use and infections in nursing homes. Tidsskr Nor Laegeforen. 2017 Mar 7;137(5):357-361. doi: 10.4045/tidsskr.16.0621. eCollection 2017 Mar. English, Norwegian. PMID 28272565
- [Derived] Heltveit-Olsen SR, Arnljots ES, Sundvall PD, Gunnarsson R, Kowalczyk A, Godycki-Cwirko M, Platteel TN, Groen WG, Lithen SS, Sundvall S, Ahren C, Grude N, Verheij TJM, Hertogh CMPM, Lindbaek M, Hoye S. Methenamine hippurate as prophylaxis for recurrent urinary tract infections in older women-a triple-blind, randomised, placebo-controlled, phase IV trial (ImpresU). Clin Microbiol Infect. 2025 Nov;31(11):1873-1879. doi: 10.1016/j.cmi.2025.07.006. Epub 2025 Jul 14. PMID 40669691
- [Derived] Heltveit-Olsen SR, Sundvall PD, Gunnarsson R, Snaebjornsson Arnljots E, Kowalczyk A, Godycki-Cwirko M, Platteel TN, Koning HAM, Groen WG, Ahren C, Grude N, Verheij TJM, Hertogh CMPM, Lindbaek M, Hoye S. Methenamine hippurate to prevent recurrent urinary tract infections in older women: protocol for a randomised, placebo-controlled trial (ImpresU). BMJ Open. 2022 Nov 1;12(11):e065217. doi: 10.1136/bmjopen-2022-065217. PMID 36319057

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04077580/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT04077580/SAP_001.pdf